CLINICAL TRIAL: NCT06246812
Title: Examining the Effects of Text Message and Competition-Based Interventions on Physical Activity, Self-Efficacy, Self-Regulation, Social Support, Incentive Motivation, and Mental Well-being Among University Students
Brief Title: Text Message and Competition-Based Interventions Among University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Collaborators: Edward Via Virginia College of Osteopathic Medicine (Other)
Responsible Party: Principal Investigator, Chenyu Zou, Principal Investigator, Auburn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-380 EX 2209
Record Dates: First submitted 2023-10-21; First posted 2024-02-07 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Physical Inactivity
Keywords: Text message; Fitness Competition; University students; Social Cognitive theory
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DFFC Group (Experimental): Students who participated in the 2022 DFFC
  Interventions: Behavioral: Deans' Fit Family Challenge
- DFFC + Text Group (Experimental): Students who participated in the 2022 DFFC and received text messages
  Interventions: Behavioral: Deans' Fit Family Challenge; Behavioral: Text message
- Control Group (No Intervention): Students who did not participate in the 2022 DFFC

INTERVENTIONS:
Behavioral: Deans' Fit Family Challenge — An annual 8-week physical activity and weight loss competition between VCOM-Auburn, AU College of Nursing, and AU Harrison School of Pharmacy
  Arms: DFFC + Text Group; DFFC Group
Behavioral: Text message — Three text messages per week to promote and motive physical activity
  Arms: DFFC + Text Group

SUMMARY:
The goal of this quasi-experimental study is to assess and compare the effectiveness of text message interventions and a competition-based intervention and evaluate participants' acceptability and experiences in university students. The main questions it aims to answer are:

1. What are the effects of text message interventions and competition-based interventions on university students' physical activity levels, self-efficacy, self-regulation, social support, incentive motivation, and mental well-being?
2. What are participants' perceptions regarding their experience with and acceptability of text message interventions and competition-based interventions?

Participants will

1. participate in a fitness competition
2. participate in a fitness competition and receive text messages
3. enroll in control group

DETAILED DESCRIPTION:
Physical activity promotes health and wellness, yet many U.S. university students are physically inactive. Text messaging and competition-based interventions have been shown to increase physical activity. The primary objectives of this study are to 1) assess and compare the effectiveness of a competition-based intervention with and without a Social Cognitive Theory-based text-messaging campaign in improving physical activity among university students, and 2) evaluate participants' acceptability and experiences of the text messaging and the competition-based interventions. In coordination with the Deans' Fit Family Challenge (DFFC; an annual physical activity and weight loss competition between Edward Via College of Osteopathic Medicine - Auburn Campus (VCOM-Auburn), Auburn University College of Nursing (AUCON), and Auburn University Harrison College of Pharmacy(HCOP), a 3-group quasi-experimental design will be employed to accomplish the study objectives. A total of 300 students will be enrolled. Students across all 3 institutions who sign up for the DFFC and enroll in this study will be randomly assigned to a competition-only group or a competition + text messaging group. The 3rd group will include students across all 3 institutions who enroll in the study but are not participating in the DFFC.

Participants will submit physical activity minutes via the "Challenge Runner" app, after initially connecting the app to their fitness tracker. All participants will be asked to complete the first anonymous survey at the beginning of the study, as well as the second anonymous survey at the conclusion of the study. Variables of interest include weekly activity minutes, self-efficacy, self-regulation, social support, incentive motivation, mental well-being, participants' acceptability and experiences, and maintenance of moderate and vigorous activity 4 weeks after DFFC. Data will be analyzed using descriptive statistics to characterize the sample and inferential statistics to analyze associations.

ELIGIBILITY:
Inclusion Criteria:

* Auburn University Harrison College of Pharmacy (HCOP), Auburn University College of Nursing (AUCON), and Edward Via College of Osteopathic Medicine - Auburn Campus (VCOM - Auburn) students
* Possess a smartphone and a fitness tracker or smartwatch
* Willingness to receive text messages

Exclusion Criteria:

* Pregnant women
* Disabilities or chronic diseases that prevent them from being physically active

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-12-11 (Actual)

PRIMARY OUTCOMES:
Minutes of weekly moderate to vigorous physical activity | week 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
  Self-reported via the ChallengeRunner online platform

SECONDARY OUTCOMES:
Self Efficacy assessed by 9-item Exercise Self Efficacy Scale | week 0 and 8
  The Self Efficacy for Exercise scale consists of nine situations (weather, boredom, pain, exercising alone, not pleasurable, too busy, feel tired, stress, depressed) that might effect participation in exercise.
Self Regulation assessed by 10-item Self-Regulation Scale | week 0 and 8
  A self-report questionnaire to assess attention control in goal pursuit.
Social Support assessed by 5-item Friend Support for Exercise Habits Scale | week 0 and 8
  Part of the Social Support for Exercise Scale developed by Sallis and colleagues.
Incentive Motivation assessed by 23-item Physical Activity Motivation Scale | week 0 and 8
  The 23-item Physical Activity Motivation Scale consists of six groups of factors: intrinsic, integrated, identified, introjected, external, and amotivation.
Mental Well-Being assessed by The World Health Organization Five Well-Being Index | week 0 and 8
  A short self-reported measure of current mental wellbeing.
Participants' Experience assessed by questionnaires | week 8
  Two multiple choice questions and two open-ended questions
Participants' Acceptability assessed by questionnaires | week 8
  Two 5-point Likert scale questions

OTHER OUTCOMES:
Race | week 0
Ethnicity | week 0
Gender | week 0
Age | week 0
Health Literacy assessed by Brief Health Literacy Screening Tool | week 0
  The BRIEF consists of the following questions: (1) How often do you have someone help you read hospital materials?"; (2) How confident are you filling out medical forms by yourself?"; (3) "How often do you have problems learning about your medical condition because of difficulty understanding written information?"; and (4) "How often do you have a problem understanding what is told to you about your medical condition?"

CONTACTS AND LOCATIONS:
Overall Officials: Brent I Fox, Study Director — Auburn University
Locations (2):
- United States (2):
  - Auburn University, Auburn, Alabama
  - Edward Via College of Osteopathic Medicine - Auburn Campus, Auburn, Alabama

REFERENCES:
- [Background] Rovniak LS, Anderson ES, Winett RA, Stephens RS. Social cognitive determinants of physical activity in young adults: a prospective structural equation analysis. Ann Behav Med. 2002 Spring;24(2):149-56. doi: 10.1207/S15324796ABM2402_12. PMID 12054320
- [Background] Farren GL, Zhang T, Martin SB, Thomas KT. Factors related to meeting physical activity guidelines in active college students: A social cognitive perspective. J Am Coll Health. 2017 Jan;65(1):10-21. doi: 10.1080/07448481.2016.1229320. Epub 2016 Sep 3. PMID 27593500
- [Background] Feng D, Zhang Y. College Students' Knowledge, attitudes, and practices regarding body posture: A cross-sectional survey--Taking a university in Wuhu City as an example. Prev Med Rep. 2023 Sep 16;36:102422. doi: 10.1016/j.pmedr.2023.102422. eCollection 2023 Dec. PMID 37736309
- [Background] Jeftic I, Furzer B, Dimmock JA, Wright K, Budden T, Boyd C, Simpson A, Rosenberg M, Sabiston CM, deJonge M, Jackson B. The Stride program: Feasibility and pre-to-post program change of an exercise service for university students experiencing mental distress. Psychol Sport Exerc. 2023 Nov;69:102507. doi: 10.1016/j.psychsport.2023.102507. Epub 2023 Aug 16. PMID 37665942